CLINICAL TRIAL: NCT01864629
Title: Optimizing Postpartum Contraception in Women With Preterm Births
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB_00061119
Record Dates: First submitted 2013-05-11; First posted 2013-05-29 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Method of Contraception; Preterm Birth Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Contraception after preterm birth (Other): Intervention name: Focused contraception counseling This intervention will be provided to those randomized to the intervention group only. This counseling will follow a pre-written, structured script describing all contraceptive methods in rank order starting with most effective to least effective in preventing unplanned pregnancy.
  Interventions: Behavioral: Focused contraception counseling
- Control Group (No Intervention): Participants will receive the standard postpartum contraception counseling that is received by all patients who deliver at our institution.

INTERVENTIONS:
Behavioral: Focused contraception counseling — This intervention will be provided to those randomized to the intervention group only. This counseling will follow a pre-written, structured script describing all contraceptive methods in rank order starting with most effective to least effective in preventing unplanned pregnancy.
  Arms: Contraception after preterm birth

SUMMARY:
The purpose of this study is to examine the effectiveness of focused family planning counseling on the uptake and continuation of highly effective contraceptive methods (defined as the intrauterine device, implant, and both male and female sterilization methods including vasectomy, tubal ligation and Essure) during the postpartum period in women who have recently experienced a preterm delivery.

The investigators hypothesize that women with a recent preterm birth (PTB) will be more likely to initiate and continue using a highly effective method of contraception when provided with focused family planning counseling.

ELIGIBILITY:
Inclusion Criteria:

* Women who deliver a premature infant that is between the gestational ages of 24 weeks 0 days and 36 weeks 6 days at our institution.

Exclusion Criteria:

* Women who have delivered via cesarean section and have also had a sterilization procedure at the time of the cesarean section.

Ages: 14 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 134 (Actual)
Dates: Start 2013-04; Primary Completion 2014-10 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Use of highly effective method | Three months

SECONDARY OUTCOMES:
Pregnancy outcomes | 12 months, 18 months, 24 months, 36 months
Use of highly effective method | 12 months, 24 months, 36 months

CONTACTS AND LOCATIONS:
Overall Officials: David K Turok, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah Hospital, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No